CLINICAL TRIAL: NCT00903201
Title: A Randomized, Double Blind, Parallel Group, Placebo Controlled 28 Day Study to Investigate the Safety, Tolerability and Pharmacodynamics of SB-656933 in Patients With Cystic Fibrosis.
Brief Title: 28 Day Repeat Dose in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110399; NCT01051453 (obsolete NCT alias)
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-08

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — SB 656933

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment A (Experimental): 20 mg of SB656933
  Interventions: Drug: SB656933
- Treatment B (Experimental): 50 mg of SB656933
  Interventions: Drug: SB656933
- Placebo (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB656933 — 20 mg
  Arms: Treatment A
Drug: SB656933 — 50mg
  Arms: Treatment B
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the safety, tolerability and pharmacodynamics of SB656933 in patients that have cystic fibrosis

DETAILED DESCRIPTION:
This proof of mechanism study aims to evaluate the safety, tolerability and pharmacodynamics of SB-656933 following 28 days of daily administration of 20 and 50 mg SB-656933 in patients with CF compared to placebo. The primary endpoints of the study will be the effect of SB-656933 on safety and tolerability (adverse events, vital signs, clinical laboratory assessments, 12-lead electrocardiograms, and urinalysis) following 28 days of dosing. Secondary endpoints will include levels of neutrophil elastase in induced sputum and other sputum markers of inflammation (e.g. myeloperoxidase, total protein), induced sputum cells (i.e. total sputum neutrophil counts, percent sputum neutrophils) and sputum microbiology. Other assessments will include lung function measurements (spirometry); serum and plasma markers of inflammation (e.g. fibrinogen, CC-16, CRP, MMP8, MMP9, SP-D, and CXCL-8), quality of life questionnaire, and population pharmacokinetics parameters of SB-656933

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF based on the following: sweat chloride > 60 mEq/L and/or genotype with 2 identifiable mutations consistent with CF; (ΔF508 homozygote, or ΔF508 heterozygote with a second allele known to cause the disease, or two alleles known to cause a class I, II, or III mutation) and one or more clinical features consistent with CF.
* Male and female subjects aged ≥18 years of age
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until one week after the last dose.
* Patients are non-smokers or former smokers by history. Former smokers will be defined as those who have not smoked for ≥6 months. Subjects who only use chewing tobacco products may be enrolled at the discretion of the Investigator and after consultation with the GSK medical monitor.
* In the judgement of the investigator the patient is clinically stable with no change in symptoms or medication, no admissions to hospital, and no intravenous antibiotic therapy for at least 1 month prior to dosing.
* Able to perform lung function tests reliably.
* FEV1 >40% and <110% predicted.
* Excluding periods of exacerbation, FEV1 has not decreased by >15% over the past 12 months
* Clinically colonized by a bacterial organism commonly seen in cystic fibrosis other than Burkholderia cepacia (i.e. Pseudomonas spp., Staphylococcus aureus, Stenotrophomonas, B. Gladioli) as evidenced by identification in sputum culture within the past year. To be eligible a CF patient must have colonization of at least one typical CF organism.
* To be eligible, female patients must have a negative pregnancy test (urine or serum) and not be nursing at screening or prior to dosing.
* Subjects must have a QTcB or QTcF < 450 msec at screening as determined by the investigators review.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within twice (2x) the upper limit of normal at screening and bilirubin within 1.25x ULN at screening. AST, ALT, alkaline phosphatase and bilirubin >2.0 xULN (isolated bilirubin >2.0xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Male subjects must agree to use one of the contraception methods listed in Section 8.1.2. This criterion must be followed from the time of the first dose of study medication until one week after the last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination, or ECG, that is not associated with cystic fibrosis.
* Neutrophil count <1.5x109 /L
* In the judgment of the PI, the patient:
* suffers from clinically unstable pancreatic function
* has clinically significant weight loss( ≥5% after a previously stable period).
* has recent change in pancreatic enzyme requirements in the past 2 months.
* Recent viral infection (within 4 weeks of dosing), with or without steroid or antibiotic treatment. Presumed viral infection will be determined according to the judgment of the Investigator and no specific testing for virus will be required.
* Subjects unable to produce a technically acceptable sputum sample.
* Clinically significant hepatic impairment
* Evidence of cirrhosis
* Patients with elevated INR that is due to suspected vitamin K deficiency may be enrolled at the discretion of the Investigator and after consultation with the GSK medical monitor
* Blood pressure persistently >155/95 mmHg at screening.
* Positive HIV, Hepatitis B surface antigen or Hepatitis C antibody at screening.
* History of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits) within 6 months of screening.
* Urinary cotinine levels indicative of smoking.
* Use of oral or parenteral corticosteroids within 4 weeks of screening; regular use (>3 x/wk) of high dose NSAIDS (e.g. >1.6g ibuprofen/day on a regular basis), within 4 weeks of screening.
* Colonization with Burkholderia cepacia
* Subjects currently being treated for mycobacterial infection
* Subjects with presumed active Allergic Bronchopulmonary Aspergillosis (ABPA)
* Subjects who have newly started therapy with azithromycin within the past 3 months.
* In the judgment of the investigator, clinically significant hemoptysis (> 30 cc per episode) within the last 6 months
* Donation of blood in excess of 500 mL within a 56-day period prior to dosing
* Participation in a trial with any drug within 30 days or 5 half-lives (whichever is longer), or participation in a trial with a new chemical entity within 2 months prior to first dose of current study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, and cannabinoids. Subjects who use benzodiazepines or other anxiolytic on a regular basis can be included at the discretion of the investigator and in consultation with the GSK medical monitor
* Patients may not be on an inhaled antibiotic during the study (i.e. must be an "off-TOBI" month; cessation of TOBI or other inhaled antibiotics commences from one week prior to dosing until final PK draw). Patients on maintenance therapy with hypertonic saline solution or inhaled DNase may continue these therapies.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2009-09-28 (Actual); Primary Completion 2010-12-29 (Actual); Study Completion 2010-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- United States (17):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Colchester, Vermont
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (5):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Reims
- Germany (6):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Israel (3):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Petah Tikva

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Moss RB, Mistry SJ, Konstan MW, Pilewski JM, Kerem E, Tal-Singer R, Lazaar AL; CF2110399 Investigators. Safety and early treatment effects of the CXCR2 antagonist SB-656933 in patients with cystic fibrosis. J Cyst Fibros. 2013 May;12(3):241-8. doi: 10.1016/j.jcf.2012.08.016. Epub 2012 Sep 17. PMID 22995323
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 110399 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110399 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110399 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110399 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110399 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110399 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110399 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 16 centers in the United States of America, 6 centers in Germany, 5 centers in France, 3 centers in Israel and 1 center in Canada from 28 September 2009 to 29 December 2010.
Pre-assignment Details: Participants were screened for a period of 28 days and at that time their eligibility for study inclusion was assessed. A total of 146 participants with cystic fibrosis were randomized to receive either 20 mg, 50 mg SB656933 or placebo orally for 28 days.
Groups:
- Placebo: Eligible participants received SB656933 matching placebo tablets via oral route, two tablets each morning, for a total of 28 days.
- SB656933 20 mg: Eligible participants received SB656933 20 milligrams (mg) tablets (two tablets of 10 mg each, every morning) via oral route, for a total of 28 days.
- SB656933 50 mg: Eligible participants received two tablets (one tablet of SB656933 50 mg and one SB656933 matching placebo tablet) each morning, via oral route, for a total of 28 days.
Period: Overall Study
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Started | 61 | 44 | 41
Completed | 56 | 38 | 39
Not Completed | 5 | 6 | 2
Not completed — Adverse Event | 1 | 4 | 0
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SB656933 20 mg: Eligible participants received SB656933 20 mg tablets (two tablets of 10 mg each, every morning) via oral route, for a total of 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg | Total
Number analyzed (Participants) | 61 | 44 | 41 | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.5 (8.41) | 32.9 (11.65) | 31.3 (12.12) | 31.0 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 17 | 55
  Male | 39 | 28 | 24 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 59 | 43 | 41 | 143
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to Follow-up (up to 42 days)
Population: All Subjects population which comprised of all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Participants
  AE | 46 | 32 | 32
  SAE | 2 | 2 | 2

2. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance
Description: Vital signs included heart rate, systolic and diastolic blood pressure and body temperature. Prior to vital signs all participants rested for at least five minutes in the seated, semi-supine, or supine position. The choice of position was kept constant for the duration of the study. Any results falling outside the normal range were repeated at the discretion of the Investigator. Potential clinical concern range for systolic blood pressure: <85 and >160 millimeter of mercury (mmHg), for diastolic: <45 and >100 mmHg and heart rate: <40 and >110 beats per minute. Number of participants with vital signs of potential clinical importance are presented.
Time Frame: Up to Follow-up (up to 42 days)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Hematology Abnormalities of Potential Clinical Importance
Description: Hematology parameters were reviewed prior to participants receiving first dose of study medication. The potential clinical concern range for hematology parameters were: Red blood cell (RBC) count (low: < 3.72 * 10^12/Liters (L) and high: > 6.313 * 10^12/L), lymphocytes (low: < 0.8 gigacells/L), hematocrit (low: > 0.075 ratio change from Baseline and high: > 0.54 ratio), mean cell hemoglobin (MCH) (low: < 23.8 picograms (pg) and high: > 39.6 pg), mean cell volume (MCV) (low: <73 femtoliters (FL) and high: >110 FL), platelet count (low: < 100 gigacells/L and high: > 550 gigacells/L), white blood cell (WBC) count (low: < 3 gigacells/L and high: > 20 gigacells/L) and eosinophils (high: > 1 gigacells/L). Only those parameters for which at least one value of potential clinical concern was reported are summarized. Number of participants with hematology abnormalities of potential clinical importance are presented.
Time Frame: Up to Follow-up (up to 42 days)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Participants
  Low RBC | 2 | 1 | 0
  High RBC | 1 | 0 | 0
  Low lymphocytes | 2 | 0 | 1
  Low MCH | 2 | 0 | 0
  Low MCV | 2 | 0 | 0
  Low Hematocrit | 1 | 0 | 0
  High platelet count | 1 | 0 | 0
  High WBC | 1 | 0 | 0
  High Eosinophils | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance
Description: The potential clinical concern range for clinical chemistry parameters were: glucose (low: < 2.8 millimole [mmol]/L and high: > 9.4 mmol/L), creatine kinase (high: > 3 * upper limit of normal units [ULN]/L), phosphorous, inorganic (low: < 0.8 mmol/L and high: > 1.6 mmol/L), total bilirubin (high: ≥ 1.5 * ULN micromole [μmol]/L), uric acid (low: < 41.636 μmol/L and high: > 582.904 μmol/L), alkaline phosphatase (ALP) (high: ≥ 2 * ULN international units [IU/L]/L), gamma glutamyl transpeptidase (GGT) (high: ≥ 110 IU/L), carbon dioxide content (low: < 18 mmol/L and high: > 32 mmol/L), direct bilirubin (high: > 1.5 * ULN μmol/L), potassium (low: < 3.0 mmol/L and high: > 5.5 mmol/L) and aspartate aminotransferase (AST) (high: ≥ 3* ULN IU/L). Only those parameters for which at least one value of potential clinical concern was reported are summarized. Number of participants with clinical chemistry abnormalities of potential clinical importance.
Time Frame: Up to Follow-up (up to 42 days)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Participants
  High Glucose | 10 | 12 | 7
  Low Glucose | 3 | 4 | 3
  High Creatine Kinase | 2 | 0 | 2
  High Phosphorous, inorganic | 4 | 0 | 2
  Low Phosphorous, inorganic | 2 | 6 | 4
  High Total Bilirubin | 2 | 2 | 0
  High Uric acid | 4 | 2 | 4
  High ALP | 3 | 1 | 2
  High GGT | 3 | 1 | 2
  Low CO2 | 3 | 3 | 4
  High Direct Bilirubin | 1 | 0 | 0
  High Potassium | 0 | 1 | 1
  High AST | 0 | 0 | 1

5. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Prior to ECG recordings, all participants rested for at least 5 minutes in the seated, semi-supine, or supine position. The choice of position was kept constant for the duration of the study. Participants avoided hot and cold food for at least 30 minutes prior to an ECG measurement. Any results falling outside normal range were repeated at the discretion of the Investigator. ECG Baseline values taken within 2.5 hours prior to first dose were calculated using the mean value of triplicate pre-dose readings. Triplicate readings were taken at least five minutes apart. Participants agreed to abstain from hot and cold drinks and food prior to an ECG measurement. ECG machine calculated heart rate and measured PR, QRS, QT, and QT corrected by Bazett's formula (QTcB), QT corrected by Fridericia's formula (QTcF) intervals. Number of participants with abnormal (not clinically significant [NCS] and clinically significant [CS]) electrocardiogram (ECG) findings are presented.
Time Frame: Up to Follow-up (up to 42 days)
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Participants
  Day 1/Pre-dose 1, Abnormal-NCS | 9 | 1 | 8
  Day 1/Pre-dose 1, Abnormal-CS | 0 | 0 | 0
  Day 1/Pre-dose 2, Abnormal-NCS: number analyzed (Participants) | 60 | 43 | 40
  Day 1/Pre-dose 2, Abnormal-NCS | 9 | 0 | 6
  Day 1/Pre-dose 2, Abnormal-CS: number analyzed (Participants) | 60 | 43 | 40
  Day 1/Pre-dose 2, Abnormal-CS | 0 | 0 | 0
  Day 1/Pre-dose 3, Abnormal-NCS: number analyzed (Participants) | 60 | 43 | 40
  Day 1/Pre-dose 3, Abnormal-NCS | 9 | 0 | 6
  Day 1/Pre-dose 3, Abnormal-CS: number analyzed (Participants) | 60 | 43 | 40
  Day 1/Pre-dose 3, Abnormal-CS | 0 | 0 | 0
  Day 14/Pre-dose 1, Abnormal-NCS: number analyzed (Participants) | 59 | 41 | 41
  Day 14/Pre-dose 1, Abnormal-NCS | 6 | 2 | 6
  Day 14/Pre-dose 1, Abnormal-CS: number analyzed (Participants) | 59 | 41 | 41
  Day 14/Pre-dose 1, Abnormal-CS | 0 | 0 | 0
  Day 28/Pre-dose 1, Abnormal-NCS: number analyzed (Participants) | 58 | 38 | 39
  Day 28/Pre-dose 1, Abnormal-NCS | 10 | 3 | 3
  Day 28/Pre-dose 1, Abnormal-CS: number analyzed (Participants) | 58 | 38 | 39
  Day 28/Pre-dose 1, Abnormal-CS | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Cystic Fibrosis (CF) Exacerbation
Description: CF is one of the most common, lethal, autosomal recessive disease characterized by airway obstruction, bronchiectasis and infection, and exocrine pancreatic insufficiency. Number of participants with CF exacerbation are presented.
Time Frame: Day 1 to Day 42
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Participants | 8 | 4 | 7

7. Secondary Outcome: Number of Participants With Pseudomonas Aeruginosa and Staphylococcus Aureus Count in Sputum
Description: Bacterial colony count of both Pseudomonas aeruginosa and Staphylococcus aureus in sputum were performed. Participants were graded as no bacteria in sputum, 1+, 2+, 3+ and 4+, which indicated proportional concentration of Pseudomonas aeruginosa and Staphylococcus aureus in sputum, where no bacteria indicated there was no bacteria in sputum, 1+ indicated slightly positive and 4+ indicated highly positive. Higher grades (4+) indicated worst outcomes (highly infected sputum). Number of participants with Pseudomonas aeruginosa and staphylococcus aureus count in sputum are presented.
Time Frame: Day 1 and Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Participants
  Pseudomonas aeruginosa: Day 1, No bacteria | 41 | 26 | 26
  Pseudomonas aeruginosa: Day 1, 1+ | 0 | 0 | 4
  Pseudomonas aeruginosa: Day 1, 2+ | 8 | 6 | 3
  Pseudomonas aeruginosa: Day 1, 3+ | 8 | 3 | 5
  Pseudomonas aeruginosa: Day 1, 4+ | 1 | 3 | 0
  Pseudomonas aeruginosa: Day 1, No sample | 3 | 6 | 3
  Pseudomonas aeruginosa: Day 28, No bacteria | 39 | 20 | 29
  Pseudomonas aeruginosa: Day 28, 1+ | 0 | 1 | 0
  Pseudomonas aeruginosa: Day 28, 2+ | 8 | 8 | 3
  Pseudomonas aeruginosa: Day 28, 3+ | 5 | 5 | 2
  Pseudomonas aeruginosa: Day 28, 4+ | 2 | 1 | 2
  Pseudomonas aeruginosa: Day 28, No sample | 7 | 9 | 5
  Staphylococcus aureus: Day 1, No bacteria | 32 | 20 | 20
  Staphylococcus aureus: Day 1, 1+ | 7 | 4 | 3
  Staphylococcus aureus: Day 1, 2+ | 7 | 7 | 1
  Staphylococcus aureus: Day 1, 3+ | 7 | 3 | 8
  Staphylococcus aureus: Day 1, 4+ | 5 | 4 | 6
  Staphylococcus aureus: Day 1, No sample | 3 | 6 | 3
  Staphylococcus aureus: Day 28, No bacteria | 35 | 18 | 17
  Staphylococcus aureus: Day 28, 1+ | 1 | 3 | 4
  Staphylococcus aureus: Day 28, 2+ | 6 | 3 | 5
  Staphylococcus aureus: Day 28, 3+ | 10 | 10 | 4
  Staphylococcus aureus: Day 28, 4+ | 2 | 1 | 6
  Staphylococcus aureus: Day 28, No sample | 7 | 9 | 5

8. Secondary Outcome: Induced Sputum Neutrophil Number
Description: Sputum samples were taken after bronchodilation and number of neutrophils in induced sputum were reported.
Time Frame: Day 28
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 10^4 cells/gram
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 49 | 35 | 34
10^4 cells/gram | 8640.0 (124.4) | 10496.2 (117.5) | 6265.4 (202.0)

9. Secondary Outcome: Induced Sputum Neutrophil Percentage
Description: Sputum samples were taken after bronchodilation and percentage of neutrophils in induced sputum are presented.
Time Frame: Day 28
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of neutrophil cells
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 49 | 35 | 34
Percentage of neutrophil cells | 91.72 (4.268) | 91.16 (4.614) | 90.83 (7.860)

10. Secondary Outcome: Induced Sputum Inflammatory Markers-Myeloperoxidase and Neutrophil Elastase
Description: Sputum samples were taken after bronchodilation. Mean induced sputum inflammatory markers namely Myeloperoxidase and neutrophil elastase are presented.
Time Frame: Day 28
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/microgram
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Nanogram/microgram
  Myeloperoxidase: number analyzed (Participants) | 52 | 37 | 37
  Myeloperoxidase | 23.2814 (78.8) | 23.4163 (62.3) | 19.6353 (104.7)
  Neutrophil elastase: number analyzed (Participants) | 49 | 34 | 35
  Neutrophil elastase | 11.2362 (276.4) | 16.5978 (113.3) | 8.7876 (361.5)

11. Secondary Outcome: Serum and Plasma Markers of Inflammation- Clara Cell Secretory Protein (CC-16) and CXCL8 (Interleukin-8 [IL-8])
Description: Blood samples intended for CC-16 and CXCL8 were collected in 5.0 milliliter (mL) serum separator goldtopped blood collection tubes, then immediately mixed by gentle inversion 10 times. The samples were permitted to coagulate for 30 to 60 minutes before centrifugation at 1600 g for 15 minutes. Two 0.75 mL aliquots of serum supernatant were transferred separately into two Sarstedt tubes and frozen at -70 degree Celsius (°C). Plasma samples intended for CC-16 and CXCL8 were centrally analyzed using a commercial test kit based on enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Day 14 and Day 28
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Picogram per milliliter
  CC-16: Day 14: number analyzed (Participants) | 59 | 41 | 41
  CC-16: Day 14 | 5148.2 (55.0) | 5507.8 (56.3) | 5610.4 (46.9)
  CC-16: Day 28: number analyzed (Participants) | 56 | 37 | 37
  CC-16: Day 28 | 5497.6 (59.2) | 5818.1 (63.7) | 6012.9 (49.7)
  CXCL8 (IL-8): Day 14: number analyzed (Participants) | 59 | 41 | 41
  CXCL8 (IL-8): Day 14 | 12.09 (54.6) | 15.75 (57.6) | 23.24 (68.4)
  CXCL8 (IL-8): Day 28: number analyzed (Participants) | 56 | 37 | 37
  CXCL8 (IL-8): Day 28 | 10.89 (66.9) | 15.68 (42.0) | 19.98 (53.8)

12. Secondary Outcome: Serum and Plasma Markers of Inflammation- C-reactive Protein (CRP)
Description: Blood samples intended for C-Reactive Protein (CRP) analysis were collected in 4.0 mL plain red-topped blood collection tubes. The samples were permitted to coagulate for 30 to 60 minutes before centrifugation at 1600 gram (g) for 15 minutes. A 1 mL volume of serum supernatant was transferred via pipette into a Nunc tube and stored at room temperature. Central analysis of CRP in serum samples was measured via fixed time nephelometry on the Behring Nephelometer II.
Time Frame: Day 14 and Day 28
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram per liter
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Milligram per liter
  Day 14: number analyzed (Participants) | 58 | 41 | 41
  Day 14 | 3.37 (229.0) | 2.72 (250.2) | 5.44 (204.2)
  Day 28: number analyzed (Participants) | 58 | 38 | 39
  Day 28 | 3.29 (231.2) | 2.88 (231.1) | 5.67 (187.3)

13. Secondary Outcome: Serum and Plasma Markers of Inflammation- Fibrinogen
Description: Blood samples intended for fibrinogen analysis were collected in 4.5 mL 3.2 % sodium citrate blue-topped blood collection tubes, then immediately mixed by gentle inversion eight to ten times. Each sample was centrifuged at 1600 g for 15 minutes. A 1 mL volume of plasma supernatant was transferred via pipette into a Nunc tube, frozen at -20°C. Central analysis of fibrinogen in plasma samples was completed via photometric clot detection with automatic sample preparation.
Time Frame: Day 14 and Day 28
Population: All Subjects Population. Only those participants available at the specified time points were analyzed. One participant in the SB656933 20 mg arm had a fibrinogen reading on Day 14. This was not a planned visit schedule, therefore, fibrinogen levels were not analyzed for the placebo arm and SB656933 50 mg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Gram per liter
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Gram per liter
  Day 14: number analyzed (Participants) | 0 | 1 | 0
  Day 14 |  | 2.240 (NA) — Single participant |
  Day 28: number analyzed (Participants) | 54 | 36 | 37
  Day 28 | 3.442 (24.1) | 3.259 (25.5) | 3.717 (20.5)

14. Secondary Outcome: Serum and Plasma Markers of Inflammation- Matrix Metalloproteinase-8 (MMP8), Matrix Metalloproteinase-9 (MMP9) and Surfactant Protein D (SP-D)
Description: Blood samples intended for MMP-8 and MMP-9 analyses were collected in 4.0 mL lithium heparin greentopped collection tubes, then immediately mixed by gentle inversion five times. The samples were centrifuged at 1800 g for 15 minutes within 30 minutes of collection. A 2 mL volume of supernatant was transferred into a Sarstedt tube and subsequently centrifuged at 10000 g for 10 minutes at 2 to 8°C for complete platelet removal. A 1 mL volume of plasma supernatant was transferred into a Sarstedt tube and frozen at -70°C. Blood samples intended for SP-D were collected in 5.0 mL serum separator goldtopped blood collection tubes, then immediately mixed by gentle inversion 10 times. The samples were permitted to coagulate for 30 to 60 minutes before centrifugation at 1600 g for 15 minutes. Two 0.75 mL aliquots of serum supernatant were transferred separately into two Sarstedt tubes and frozen at -70°C. Plasma samples were centrally analyzed using a commercial test kit based on ELISA method.
Time Frame: Day 14 and Day 28
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
Nanogram per milliliter
  MMP8: Day 14: number analyzed (Participants) | 59 | 39 | 41
  MMP8: Day 14 | 11.407 (109.0) | 8.808 (136.5) | 7.626 (143.3)
  MMP8: Day 28: number analyzed (Participants) | 56 | 36 | 37
  MMP8: Day 28 | 10.136 (113.2) | 9.188 (137.7) | 9.043 (119.0)
  MMP9: Day 14: number analyzed (Participants) | 59 | 39 | 41
  MMP9: Day 14 | 122.31 (104.8) | 107.40 (81.6) | 85.72 (93.4)
  MMP9: Day 28: number analyzed (Participants) | 56 | 36 | 37
  MMP9: Day 28 | 116.31 (87.1) | 115.32 (89.4) | 106.60 (107.4)
  SP-D: Day 14: number analyzed (Participants) | 59 | 41 | 41
  SP-D: Day 14 | 10.707 (76.8) | 9.735 (88.3) | 9.367 (74.2)
  SP-D: Day 28: number analyzed (Participants) | 56 | 37 | 37
  SP-D: Day 28 | 10.428 (80.6) | 10.037 (90.7) | 10.042 (67.9)

15. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) and Forced Vital Capacity (FVC)
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FVC is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (Day 1) to Day 14 and Day 28
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (90% Confidence Interval); unit: L
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 61 | 44 | 41
L
  FEV1: Day 14: number analyzed (Participants) | 58 | 40 | 41
  FEV1: Day 14 | 0.040 [-0.020 to 0.101] | -0.065 [-0.138 to 0.007] | -0.036 [-0.108 to 0.036]
  FEV1: Day 28: number analyzed (Participants) | 54 | 37 | 39
  FEV1: Day 28 | 0.031 [-0.026 to 0.087] | -0.031 [-0.099 to 0.037] | -0.013 [-0.080 to 0.054]
  FVC: Day 14: number analyzed (Participants) | 58 | 40 | 41
  FVC: Day 14 | -0.005 [-0.069 to 0.058] | -0.072 [-0.148 to 0.005] | -0.017 [-0.092 to 0.059]
  FVC: Day 28: number analyzed (Participants) | 54 | 37 | 39
  FVC: Day 28 | -0.018 [-0.085 to 0.048] | -0.021 [-0.101 to 0.059] | 0.022 [-0.056 to 0.101]

16. Secondary Outcome: Area Under the Plasma Drug Concentration (AUC) Versus Time Curve: AUC From Time Zero (Pre-dose) to Four Hours Post Dose (AUC[0-4]) and AUC From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC[0-t])
Description: Blood samples were taken via an indwelling cannula (or by direct venepuncture), collected into a 3.0 mL Ethylenediaminetetraacetic acid (EDTA) lavender-topped collection tube, immediately mixed by gentle inversion ten times, then placed on water ice. The samples were centrifuged at 1600 g for 15 minutes at 4°C for 10 minutes. Supernatant plasma was transferred to a 1.8 mL Nunc tube and frozen at -20°C.
Time Frame: Day 1: pre-dose, 0.5, 1, 2, 4 and 8 hours post-dose and Day 28: pre-dose, 1 and 4 hours
Population: PK Population which comprised of all participants in the 'All Subjects' population for whom a pharmacokinetic sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram * hour/milliliter (ng*h/mL)
Arm/Group | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 44 | 41
Nanogram * hour/milliliter (ng*h/mL)
  AUC(0-4): Day 1 | 747.1 (63.8) | 2227.6 (44.8)
  AUC(0-4): Day 28: number analyzed (Participants) | 38 | 39
  AUC(0-4): Day 28 | 592.3 (93.1) | 1906.8 (85.1)
  AUC(0-t): Day 1 | 1272.5 (42.6) | 3537.6 (45.0)
  AUC(0-t): Day 28: number analyzed (Participants) | 38 | 39
  AUC(0-t): Day 28 | 592.3 (93.1) | 1906.8 (85.1)

17. Secondary Outcome: Maximum Observed Plasma Drug Concentration (Cmax)
Description: Blood samples were taken via an indwelling cannula (or by direct venepuncture), collected into a 3.0 mL EDTA lavender-topped collection tube, immediately mixed by gentle inversion ten times, then placed on water ice. The samples were centrifuged at 1600 g for 15 minutes at 4°C for 10 minutes. Supernatant plasma was transferred to a 1.8 mL Nunc tube and frozen at -20°C.
Time Frame: Day 1: pre-dose, 0.5, 1, 2, 4 and 8 hours post-dose and Day 28: pre-dose, 1 and 4 hours
Population: PK population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 44 | 41
Nanogram per milliliter
  Day 1 | 342.89 (53.6) | 967.78 (54.3)
  Day 28: number analyzed (Participants) | 38 | 39
  Day 28 | 222.86 (122.4) | 778.04 (65.2)

18. Secondary Outcome: Time to Maximum Observed Plasma Drug Concentration (Tmax)
Description: as for outcome 17
Time Frame: Day 1: pre-dose, 0.5, 1, 2, 4 and 8 hours post-dose and Day 28: pre-dose, 1 and 4 hours
Population: PK population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | SB656933 20 mg | SB656933 50 mg
Number analyzed (Participants) | 44 | 41
Hour
  Day 1 | 1.9398 [0.500 to 4.000] | 1.7362 [0.500 to 4.250]
  Day 28: number analyzed (Participants) | 38 | 39
  Day 28 | 2.1101 [0.967 to 4.083] | 1.8449 [0.950 to 4.000]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAE) and non-serious adverse events (nSAE) were collected from the first administration of study medication (Day 1) until the final follow up visit (Day 42, Visit 6).
Description: SAE and nSAE are reported for all subjects population which comprised of all participants who received at least one dose of study medication.
Arm/Group | Placebo | SB656933 20 mg | SB656933 50 mg
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/44 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/61 | 2/44 | 2/41
Other Adverse Events (participants affected / at risk) | 33/61 | 28/44 | 22/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | SB656933 20 mg (N=44) | SB656933 50 mg (N=41)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | SB656933 20 mg (N=44) | SB656933 50 mg (N=41)
Headache (Nervous system disorders) | 16 | 13 | 7
Dizziness (Nervous system disorders) | 2 | 3 | 1
Sinus headache (Nervous system disorders) | 0 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 7
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Chest discomfort (General disorders) | 5 | 3 | 5
Fatigue (General disorders) | 5 | 3 | 1
Pyrexia (General disorders) | 0 | 4 | 2
Irritability (General disorders) | 0 | 3 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 | 3 | 5
Nasopharyngitis (Infections and infestations) | 3 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 0
Pulmonary function test decreased (Investigations) | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.